CLINICAL TRIAL: NCT03495063
Title: Comparison of Synthetic and Natural Caffeine on Hemodynamic Parameters in Young, Healthy Volunteers: A Randomized, Double Blind, Crossover Study
Brief Title: Synthetic and Natural Caffeine on Hemodynamic Parameters in Young, Healthy Volunteers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to quantify caffeine
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth Tesch, PGY-1 Pharmacy Resident, David Grant U.S. Air Force Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: FDG20180007H
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Injury

STUDY DESIGN:
Intervention Model Description: This protocol uses a crossover design. The subject sample is randomized. Subjects will serve as their own controls as they will be asked to intake both the natural and synthetic caffeine at two different occasions.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural Caffeine (Experimental): Subjects will be their own control and will have repeated measures after the consumption of a drink with 400mg of natural caffeine. Blood pressure measurements will be taken at baseline, then hourly for four hours.
  Interventions: Dietary Supplement: Natural Caffeine
- Synthetic Caffeine (Experimental): Subjects will be their own control and will have repeated measures after the consumption of a drink with 400mg of synthetic caffeine. Blood pressure measurements will be taken at baseline, then hourly for four hours.
  Interventions: Dietary Supplement: Synthetic Caffeine

INTERVENTIONS:
Dietary Supplement: Natural Caffeine — Consumption of 400mg of natural caffeine
  Arms: Natural Caffeine
Dietary Supplement: Synthetic Caffeine — Consumption of 400mg of synthetic caffeine
  Arms: Synthetic Caffeine

SUMMARY:
The purpose of this study determine the difference in hemodynamic effects of synthetic and natural caffeine consumption in healthy individuals through blood pressure (central and peripheral) assessment. Participants will randomly be assigned to consume either one 8oz cup of coffee containing 400mg of caffeine (increased caffeine using concentrated coffee) or one 8oz cup of coffee-flavored drink with approximately 400mg synthetic caffeine from capsules dissolved in it.

DETAILED DESCRIPTION:
The purpose of this study is to assess the difference in effects of consuming synthetic versus natural caffeine on hemodynamic parameters in healthy subjects. This study will determine the difference in hemodynamic effects of synthetic and natural caffeine consumption in healthy individuals through blood pressure (central and peripheral) assessment. The participants in this study are healthy adults who will be introduced to a risk that may be more than they would encounter through their normal daily activities. This study seeks to add to the literature by evaluating the difference in impact of synthetic compared to natural caffeine on central blood pressure.

This protocol has the following aims:

1. Investigators hypothesize there will be a (baseline adjusted [ΔBP]) difference in BP (peripheral and central) between the natural and synthetic caffeine arms in healthy volunteers post consumption.
2. Investigators hypothesize there will be (baseline adjusted [ΔCO]) no difference in CO between the natural and synthetic caffeine arms in healthy volunteers post consumption.
3. Investigators hypothesize there will be (baseline adjusted [ΔSVR]) no difference in SVR between the natural and synthetic caffeine arms in healthy volunteers hours post consumption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Active duty military service members
* DoD beneficiaries
* Participants must be willing to refrain from caffeine use 72 hours prior to study days one and five

Exclusion Criteria:

* Cardiovascular risk factors: Heart rhythm other than normal sinus, history of atrial or ventricular arrhythmia, family history of premature sudden cardiac death before the age of 60, left ventricular hypertrophy, acute myocardial ischemia, atherosclerosis, hypertension, and palpitations. This will be determined through the questionnaire responses of the participant and thorough chart review.
* Blood pressure at initial screening appointment or at baseline on study Day One greater than 130/80 and if 130-139/80-89, FRS risk greater than 10%.
* Presence of any known medical condition, confirmed through participant interview up to the discretion of the research team. Examples of these are:
* Hypertension
* Thyroid disease
* Type 1 or 2 Diabetes Mellitus
* Recurrent headaches
* Any psychiatric condition or neurological disorder including seizures
* History of alcohol or drug abuse in the previous five years
* Ever been diagnosed or told they have or had renal or hepatic dysfunction
* Tobacco use
* Concurrent use of any medication taken in an amount greater than twice a week, to include herbal products or supplements, not to include hormonal contraceptives. If less than or equal to two days per week, the investigator will determine if the subject is to be included or excluded based on the available literature for that medication.
* Pregnant or lactating females will be excluded from participation with urine dipstick tests used to rule out pregnancy (pregnancy test performed before each treatment session, days one, five)
* All non-English speaking/writing subjects and those that do not understand the study or consent process will be excluded from the study due to unavailability of medical qualified translator at all times during the study.
* If the subject refuses to sign the informed consent document or HIPAA Authorization, they will be excluded as well.
* Allergy to any substance in the study design.
* Any other medical reason that at the discretion of the investigators would pose a risk to the health of the subject.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Peripheral systolic blood pressure | Four hours
  Two peripheral systolic blood pressure measurements will be taken prior to the consumption of the assigned study drink. Repeated peripheral systolic blood pressure readings will occur twice at each time point hourly for a period of four hours. For each measurement, participant will be asked to rest for five minutes.

SECONDARY OUTCOMES:
Change in peripheral diastolic blood pressure | Four hours
  Two peripheral diastolic blood pressure measurements will be taken prior to the consumption of the assigned study drink. Repeated peripheral diastolic blood pressure readings will occur twice at each time point hourly for a period of four hours. For each measurement, participant will be asked to rest for five minutes.
Cardiac output | Four hours
  Cardiac output will be measured prior to the consumption of assigned study drink. Repeated cardiac output readings will occur twice at each time point hourly for a period of four hours. For each measurement, participant will be asked to rest for five minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Tesch, Principal Investigator — David Grant Medical Center; Sachin A Shah, Principal Investigator — David Grant Medical Center
Locations (1):
- David Grant Medical Center, Travis Air Force Base, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fletcher EA, Lacey CS, Aaron M, Kolasa M, Occiano A, Shah SA. Randomized Controlled Trial of High-Volume Energy Drink Versus Caffeine Consumption on ECG and Hemodynamic Parameters. J Am Heart Assoc. 2017 Apr 26;6(5):e004448. doi: 10.1161/JAHA.116.004448. PMID 28446495
- [Background] Furie B, Furie BC. Mechanisms of thrombus formation. N Engl J Med. 2008 Aug 28;359(9):938-49. doi: 10.1056/NEJMra0801082. No abstract available. PMID 18753650
- [Background] Guessous I, Eap CB, Bochud M. Blood pressure in relation to coffee and caffeine consumption. Curr Hypertens Rep. 2014 Sep;16(9):468. doi: 10.1007/s11906-014-0468-2. PMID 25090963
- [Background] Hartley TR, Lovallo WR, Whitsett TL. Cardiovascular effects of caffeine in men and women. Am J Cardiol. 2004 Apr 15;93(8):1022-6. doi: 10.1016/j.amjcard.2003.12.057. PMID 15081447
- [Background] Knapik JJ, Trone DW, McGraw S, Steelman RA, Austin KG, Lieberman HR. Caffeine Use among Active Duty Navy and Marine Corps Personnel. Nutrients. 2016 Oct 9;8(10):620. doi: 10.3390/nu8100620. PMID 27735834
- [Background] Lieberman HR, Stavinoha T, McGraw S, White A, Hadden L, Marriott BP. Caffeine use among active duty US Army soldiers. J Acad Nutr Diet. 2012 Jun;112(6):902-12, 912.e1-4. doi: 10.1016/j.jand.2012.02.001. PMID 22709816
- [Background] Marik PE. Noninvasive cardiac output monitors: a state-of the-art review. J Cardiothorac Vasc Anesth. 2013 Feb;27(1):121-34. doi: 10.1053/j.jvca.2012.03.022. Epub 2012 May 19. No abstract available. PMID 22609340